CLINICAL TRIAL: NCT02420249
Title: Randomised Controlled Trial of Qigong Training Programme to Alleviate Arm Oedema, ¬Reduce Shoulder Impairment, Improve Body Balance and Quality of Life in Community-dwelling Breast Cancer Survivors
Brief Title: Qigong for Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Assistant Professor, DRPC chairperson, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201410159001
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qigong training group (Experimental): Participants assigned to the Qigong group will receive Qigong training. The Qigong training programme will be run for 3 months with two supervised 1-hour sessions per week. Participants will learn the 18 Forms of Tai Chi Internal Qigong. The training sessions will be conducted by a qualified Qigong instructor from the Natural Health Qigong Association. Participants in the control group will receive no Qigong training during the study period. They will receive an 18 Forms of Tai Chi Internal Qigong training package after the study.
  Interventions: Behavioral: Qigong training
- Control group (No Intervention): Participants in the control group will receive no Qigong training.

INTERVENTIONS:
Behavioral: Qigong training — Participants will learn the 18 Forms of Tai Chi Internal Qigong. Detailed movement and breathing descriptions of the Qigong training protocol can been found in Mak YK. 18 Forms Tai Chi Qigong [in Chinese]. 7th ed. Hong Kong: Wan Li Book Co.; 2012.
  Arms: Qigong training group

SUMMARY:
Objectives: (1) To investigate the effects of Qigong training on upper limb oedema, circulatory status, shoulder flexibility and muscular strength, body balance, and quality of life (QOL) in community-dwelling breast cancer survivors; and (2) to explore the relationship between the impairment outcomes and QOL outcomes.

Hypothesis: (1) The experimental participants will have less impairment and a better QOL after Qigong training compared with the no-training control group; and (2) the impairment parameters will be related to the QOL indexes in the Qigong participants.

Design and subjects: This will be a prospective, randomised, single-blinded controlled trial. Approximately 60 breast cancer survivors will be randomly assigned to either the Qigong training group (n~30) or control group (n~30).

Intervention: Participants in the Qigong group will receive 18 Forms of Tai Chi Internal Qigong training for 3 months with two supervised 1-hour sessions per week.

Main outcome measures: The primary outcome measures are upper limb circumference, arterial blood flow velocities and resistance index, shoulder joint passive range of motion, muscular strength (peak force) and body balance. The secondary outcome measure is quality of life as measured by the Functional Assessment of Cancer Therapy - Breast scale.

Data analysis: Data will be analysed via repeated-measures analysis of variance followed by post-hoc tests (α = 0.05).

Expected results: The investigators pilot studies produced encouraging results on the efficacy of Qigong exercise in reducing chronic breast cancer-related symptoms in survivors. Therefore, the investigators expect that participants in the Qigong group will have fewer upper limb impairments and a better quality of life after Qigong training. If the results are positive, this Qigong training regime is readily transferrable to clinical practice, and could have positive socioeconomic effects such as reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are

1. history of a breast malignancy of any stage
2. history of mastectomy or lumpectomy with or without adjuvant chemotherapy or radiotherapy
3. having completed conventional cancer treatment and medically stable
4. no known neurological deficits resulting from breast cancer treatment or other neurological disorders
5. persistent lymphoedema defined as a circumference difference greater than 2 cm at any point between the surgical upper limb and contralateral upper limb13
6. female aged 18 or above.

Exclusion Criteria:

The exclusion criteria are

1. presence of major psychiatric, neurological, musculoskeletal, cardiovascular, peripheral vascular or kidney disorder
2. receiving conventional cancer treatments such as chemotherapy or radiotherapy, medications such as diuretics or traditional Chinese medicine
3. recurrent cancer or cancer that has spread to another organ
4. participation in regular physical activity
5. prior experience of Qigong or Tai Chi
6. a smoking habit
7. pregnancy during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in upper limb circumference | Baseline (0 month) and post-intervention (3 months)
  Circumference of both arms will be measured using a cloth measuring tape.
Change in arterial resistance and blood flow velocities | Baseline (0 month) and post-intervention (3 months)
  A Doppler ultrasound machine will be used to examine the arterial blood flow velocities.
Change in shoulder flexibility | Baseline (0 month) and post-intervention (3 months)
  A universal goniometer will be used to measure the passive range of motion (ROM) of bilateral shoulder abduction and horizontal abduction.
Change in shoulder muscular strength | Baseline (0 month) and post-intervention (3 months)
  The maximum isometric muscular strength of the shoulder flexor, abductor, internal rotator and external rotator muscles will be measured bilaterally using the Lafayette Manual Muscle Test System.
Change in body balance | Baseline (0 month) and post-intervention (3 months)
  Standing balance of the participants will be measured using timed single leg standing test.

SECONDARY OUTCOMES:
Change in quality of life | Baseline (0 month) and post-intervention (3 months)
  Functional Assessment of Cancer Therapy - Breast scale version 4 will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Pokfulam, Hong Kong